CLINICAL TRIAL: NCT05691413
Title: The Safety and Efficacy of Facial Cleanser Containing Combination of Olive Oil, Virgin Coconut Oil, Butylene Glycol and Hyaluronic Acid on Skin Hydration and Skin Elasticity
Brief Title: Safety and Efficacy of Facial Cleanser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMRAMREC004-22
Record Dates: First submitted 2023-01-10; First posted 2023-01-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Aesthetic; Cosmetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Product X facial cleanser (Experimental): Participants will used Product X facial cleanser twice daily for 5 weeks
  Interventions: Other: Other: Product X facial cleanser

INTERVENTIONS:
Other: Other: Product X facial cleanser — Product X facial cleanser contain olive oil, virgin coconut oil, butylene glycol and hyaluronic acid

SUMMARY:
This study is conducted to evaluate the safety and effectiveness of facial cleanser X containing combination of olive oil, virgin coconut oil, butylene glycol and hyaluronic acid on skin hydration and skin elasticity. The study duration is 5 weeks and the skin assessment will be carried out at baseline, week 3 and week 5.The main questions this study aims to answer are:

1. The effect of product on skin hydration.
2. The effect of product on skin elasticity.
3. To observe any adverse effect occurrence with the usage of the product.

ELIGIBILITY:
Inclusion Criteria:

* Malaysia citizen
* Male and female (age 35-55 years old)

Exclusion Criteria:

* Participants who have acne which require medical treatment.
* Participants taking isotretinoin
* Participants who had undergo any cosmetic procedures such as laser & light treatment, botulinum toxin A injections and chemical peeling for the past 3 months
* Participants who are immunocompromised
* Participants with history of facial surgery

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in skin hydration from baseline and at week 3 and 5 after using facial cleanser X | Baseline, week 3 and week 5
  Skin hydration will be assessed using JANUS III skin analyzer
Change in skin elasticity from baseline and at week 3 and 5 after using facial cleanser X | Baseline, week 3 and week 5
  Skin elasticity will be assessed using JANUS III skin analyzer
Adverse effect after using facial cleanser X | Week 5
  Based on adverse effect occurrence on participants that occur during study period (5 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No